CLINICAL TRIAL: NCT01234454
Title: Risperidone Effects On Frontal And Temporal Cortical Function In Schizophrenia Patients Undergoing FMRI Cognitive Task Performance
Brief Title: Atypical Antipsychotic Treatment Effect On Brain Function In Schizophrenia Measured By FMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Aysenil Belger, Ph.D/Principal Investigator, UNC-Chapel Hill, Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RIS-USA-242
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Risperidone Treatment Group (Experimental): A two-week cross-titration phase followed randomization when patients started treatment with Risperidone in a double-blind manner and were tapered off Thiothixene. A six-week double blind active treatment period followed. Target dose was 6mg/day or highest dose tolerated.
  Interventions: Drug: Risperidone
- Olanzapine Treatment Group (Experimental): A two-week cross-titration phase followed randomization when patients started treatment with Olanzapine in a double-blind manner and were tapered off Thiothixene. A six-week double blind active treatment period followed. Target dose 20mg/day (or the highest dose tolerated) for 8 weeks, following 4 weeks of baseline Thiothixene.
  Interventions: Drug: Olanzapine
- Thiothixene (No Intervention): Subjects were first stabilized on open-label Thiothixene for four weeks, target dose 25 mg per day. Patients were then randomized to either Risperidone or Olanzapine treatment for 8 weeks.

INTERVENTIONS:
Drug: Risperidone — 6mg/day or highest dose tolerated for 8 weeks, following 4 weeks baseline treatment of Thiothixene
  Other Names: risperidol, risperidal
  Arms: Risperidone Treatment Group
Drug: Olanzapine — 20mg/day for 8 weeks, following 4 weeks of baseline Thiothixene.
  Other Names: Zydis, Zyprexa
  Arms: Olanzapine Treatment Group

SUMMARY:
The general aim is to compare the effects of typical and atypical antipsychotic medication on brain structure and function. A parallel group treatment trial will be utilized to compare the effects of the typical antipsychotic thiothixene versus the atypical antipsychotics risperidone (RIS) and olanzapine (OLZ) on brain structure and function in schizophrenia in an effort to determine the neuroanatomic basis for cognitive pathology in schizophrenia and its amelioration by atypical antipsychotic drugs.

DETAILED DESCRIPTION:
The general aim of this study was to determine the neuroanatomic basis for cognitive pathology in schizophrenia, as well as the effects of treatment with typical and atypical antipsychotics on clinical symptoms, neurocognition and brain function, as measured with function magnetic resonance imaging. Subjects underwent a randomized parallel group treatment trial that consisted of: a four-week Thiothixene treatment period, followed by randomization, two-weeks cross titration, and six-weeks of double blind treatment with Risperidone (RIS) or Olanzapine (OLZ). Twenty-three patients with schizophrenia or schizoaffective disorder and fifteen healthy control subjects were initially enrolled. Diagnosis was established with the SCID. Subjects were assessed at two time points, at baseline after four weeks of Thiothixene treatment and at follow up, after eight weeks of double-blind atypical antipsychotic treatment. Controls were assessed once. Symptom severity was assessed using the PANSS. Cognitive functions associated with frontal and temporal cortical regions were probed with a neurocognitive testing battery using standardized attention, executive function and working memory tasks. Frontal and temporal cortical function was assessed with fMRI during the performance of visual and auditory oddball tasks. The visual task oddball task consisted of identifying an infrequent square presented within a series of frequent squares. The auditory oddball task consisted of identifying an infrequent pitch-deviant target tone embedded within a series of frequent standard tones. Thirteen patients and eleven controls completed fMRI at baseline and follow-up.

The results indicated that patients treated with the typical neuroleptic Thiothixene showed significantly smaller extents of activations in superior temporal, anterior cingulate and thalamic regions as compared to control subjects during the auditory oddball task. Although treatment with atypical neuroleptics considerably reduced group differences in cortical activation between controls and patients, the current sample size proved to be insufficient to yield statistically significant group by time interactions. The percent signal change data was in the same direction, but proved to be less sensitive to group differences than the extent of activation. The group differences were not pronounced during the visual oddball task, but were in the same direction.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Schizophrenia/Schizoaffective Subjects

1. Men and women between ages of 18 to 60 inclusive, of any ethnic origin.
2. Subjects must be right handed.
3. DSM IV criteria for chronic schizophrenia or schizoaffective disorder.
4. Good physical health as determined by complete physical examination, laboratory tests, and EKG

Inclusion Criteria for Healthy Control Subjects:

1. Fifteen individuals, matched to the patient subjects on the basis of age, gender, parental SES, handedness.

Exclusion Criteria:

Exclusion Criteria for Schizophrenia/Schizoaffective Subjects

1. Previous poor response or adverse side effects to thiothixene, olanzapine or risperidone.
2. Left handedness
3. Epilepsy, HIV, or current myeloproliferative disorder
4. Current severe major depression.
5. Current or past history of Substance Dependence (except caffeine or nicotine)
6. Criteria for active Substance Abuse within past 30 days
7. Learning disability
8. Mental Retardation
9. Foreign metal objects or implants as determined by MRI safety questionnaires
10. If judged unsuitable for the study based on other medical or psychiatric condition according to the PIs best clinical judgment.
11. No depot neuroleptic within 60 days before the day of randomization.
12. Women who are pregnant or breastfeeding, and/or unwilling to take a pregnancy test.

Exclusion Criteria for Healthy Control Subjects

1. History of psychiatric disorder or current medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2002-01; Primary Completion 2005-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Assessment Procedure | Baseline, after four weeks of Thiothixine, then follow-up after 8 weeks
  Composite score derived from the neurocognitive battery used in the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) schizophrenia clinical trial and the Brief Assessment of Cognition in Schizophrenia (BACS).
fMRI activation Tasks | Baseline, after four weeks of Thiothixine, then follow-up after 8 weeks
  During MR imaging subjects performed one visual-auditory target detection task and one auditory oddball task. Subjects completed runs consisting of 160 trials with a total duration of approximately 4 min. During odd numbered runs, subjects performed a visual target detection task. During even numbered runs, subjects performed an auditory target detection task.

SECONDARY OUTCOMES:
Performance accuracy on Visual-auditory target detection task | Baseline, after four weeks of Thiothixine, then follow-up after 8 weeks
  Per fMRI activation tasks. For the visual task, subjects were asked to pay attention to a screen where two types of stimuli were displayed: 1) Standards were squares of varying size and color that comprised ~95% of trials 2) Targets were circles of varying zize and colors that were presented irriegularly on ~5% of trials. The onsets of successive Targets were separated by a minimum of 15 seconds.
Performance accuracy on Auditory oddball target detection task | baseline, after four weeks of Thiothixine, then follow-up after 8 weeks
  Per fMRI activation tasks. Subjects were asked to pay attention to attend to auditory stimuli presented at a rate of one per 500 msecs for each run. Standards were 500 msec duration 440 Hz pure tones that were presented on ~95% of trials. Frequency-deviant Target tones were 500msec duration 800 Hz pure tones presented irregularly on ~5% of trials. The onsets of successive deviant tones were separated by a minimum of 15 seconds. During both tasks subjects were instructed to press a button whenever a Target was presented. No overt or covert response was required of Standards.

CONTACTS AND LOCATIONS:
Overall Officials: AYSENIL BELGER, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Unc Psychiatry, Chapel Hill, North Carolina, United States